CLINICAL TRIAL: NCT06872437
Title: EFFICACY OF THE USUAL TREATMENT WITH INFILTRATION OF LOCAL ANAESTHETIC IN THE TREATMENT OF PUDENDAL NEURALGIA: A RANDOMISED TRIAL COMPARED WITH A PHYSIOLOGICAL SERUM
Brief Title: Evaluation of the Efficacy of Therapeutic Infiltrations of the Pudendal Nerve, Performed Under Neurostimulation on Pain, 1 Month After an Infiltration of Local Anaesthetic, in the Treatment of Pudendal Neuralgia.
Acronym: EPHI-DACI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RI-B-2021-7300-07
Record Dates: First submitted 2021-04-29; First posted 2025-03-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pudendal Neuralgia
MeSH Terms: conditions — Pudendal Neuralgia | interventions — Saline Solution; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Infiltration by injections of 6mL of lidocaine (10 mg/mL) per injection site (left ischioanal fossa, right ischioanal fossa right ischioanal fossa, coccyx)
  Interventions: Drug: Lidocaine Injectable Solution
- Saline solution (Placebo Comparator): Infiltration by injections of 6mL of saline solution per injection site (left ischio-anal fossa, right ischio-anal fossa right ischio-anal fossa, coccyx)
  Interventions: Drug: Saline Solution for Block

INTERVENTIONS:
Drug: Lidocaine Injectable Solution — Infiltration by injections of 6mL of lidocaine (10 mg/mL) per injection site (left ischioanal fossa, right ischioanal fossa right ischioanal fossa, coccyx),
  Arms: Lidocaine
Drug: Saline Solution for Block — Infiltration by injections of 6mL of saline solution per injection site (left ischio-anal fossa, right ischio-anal fossa right ischio-anal fossa, coccyx)
  Arms: Saline solution

SUMMARY:
Pudendal neuralgia (PN) is a chronic nerve compression syndrome causing neuropathic pain. Treatment includes medication, infiltration and decompressive surgery. Medicinal treatment involves the use of drugs that have proved effective in other areas, such as shingles or diabetes. There is no consensus on the molecules to be used for pudendal nerve infiltration (PNTI), and less than half of patients experience short-term relief. The only risk factor for failure is the duration of pain. Our study proposes to compare the usual treatment with a placebo, as no type of infiltration has been compared with a placebo.

DETAILED DESCRIPTION:
Like carpal tunnel syndrome, pudendal neuralgia (PN) is defined as a syndrome of chronic nerve compression (of the pudendal nerve) causing neuropathic pain.

Treatment of NP is based on 3 therapeutic strategies of increasing aggressiveness: drug treatment, infiltrations and decompressive surgery.

Drug treatment is based on the "empirical" use of drugs for neuropathic pain that have proved effective in other areas (shingles, diabetes, etc.). People with this disease are generally considered 'non-responders' to drug treatment after failure (decrease in VAS scale < 3) of at least one antidepressant and one antiepileptic drug, whose doses have been increased to the maximum possible level, or in whom a side effect has prevented the dose from being increased to the maximum authorised level.

For pudendal nerve infiltration (ITNP), there is no consensus or recommendation on which molecules to use. Most studies have used a combination of local anaesthetics and corticosteroids. However, a randomised controlled trial, researchers compare lidocaine infiltration with or without methylprednisolone. The results were not significantly different (14% vs 11%).

According to the data in the literature, less than half of patients (11% to 39%) are relieved in the short term, up to 3 months, and only about 10% (6.8% to 12.2%) are still relieved at 1 year. The only recognised risk factor for failure seems to be the duration of pain (more than 1 year). Other risk factors have been described in the literature, but only in one study and not in the others, such as gender (male or female), age (over or under 70), duration of pain (over or under 1 year), and whether the pain is bilateral or not.

In our department, patients are currently treated with lidocaine INTP under neurostimulation. Given the poor results in terms of efficacy and the strong psychological component in chronic pain pathologies, the investigators propose in this study to compare our usual treatment with placebo, since no type of infiltration has ever been compared with placebo, although this is a condition where the placebo effect is likely to be large.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* Expressed consent to participate in the study
* Affiliated or beneficiary of a social security plan
* With pudendal neuralgia (Nantes criteria "modified" Nantes criteria).
* MRI normal or without pathology explaining the pain
* Drug treatment failure as defined in the LOS, i.e., failure (VAS decrease < 3) of at least one antiepileptic drug and an antidepressant whose dosages have been to the maximum possible dosage, or in whom a side effect for whom a side effect could not allow the dose to be increased to its to its maximum allowed dose.

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* General and/or local infection (fistulous or cutaneous suppuration of the anal margin) in progress
* Known neurological pathology that may explain the pain
* Psychiatric pathology requiring a drug treatment treatment
* Anticoagulants or haemostasis disorders
* Hypersensitivity to lidocaine hydrochloride, to local anesthetics
* Recurrent porphyrias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2029-03-08 (Estimated); Study Completion 2029-03-08 (Estimated)

PRIMARY OUTCOMES:
Comparison between the two treatment arms (lidocaine vs.saline) of the rate of patients with a decrease of at least 3 points on a visual 3 points on a visual analogue pain scale (VAS) between inclusion and | between inclusion and 1 month after the first injection.

CONTACTS AND LOCATIONS:
Overall Officials: Axel EGAL, Doctor, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Hôpital Croix Saint-Simon, Paris, France

IPD SHARING:
Plan to Share IPD: No